CLINICAL TRIAL: NCT04763369
Title: Investigation of Therapeutic Efficacy and Safety of Umbilical Cord Derived Mesenchymal Stem Cells (UMSCs) for the Management of Retinitis Pigmentosa (RP)
Brief Title: Investigation of Therapeutic Efficacy and Safety of UMSCs for the Management of Retinitis Pigmentosa (RP)
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Jinnah Burn and Reconstructive Surgery Centre, Lahore (Other Government)
Collaborators: The Layton Rahmatullah Benevolent Trust (LRBT) Free Eye Hospital, Township Lahore. (Unknown); Centre of Excellence in Molecular Biology (CEMB), University of the Punjab, Lahore. (Unknown)
Responsible Party: Principal Investigator, Prof. Dr. Sheikh Riazuddin, Distinguished National Professor, Jinnah Burn and Reconstructive Surgery Centre, Lahore
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: JB&RSC-02
Record Dates: First submitted 2021-02-06; First posted 2021-02-21 (Actual); Last update posted 2021-02-21 (Actual); Status verified 2021-02

CONDITIONS: Retinitis Pigmentosa (RP)
Keywords: Retinitis pigmentosa; Stem cells treatment
MeSH Terms: conditions — Retinitis Pigmentosa

STUDY DESIGN:
Intervention Model Description: Group 1: Five (5) subjects will be treated by injecting UMSCs in sub-tenon space of eye.
  Group 2: Five (5) subjects will be treated by suprachoroidal injection of UMSCs .
  From two subjects in group 1 & 2 will not be treated 24 hrs apart. Patients will be randomized in a 1:1 ratio (Sub-tenon injection of UMSCs : Suprachoroidal injection of UMSCs).
  Note: In total, twenty five patients will be subjected to cell injection for each of group 1 & 2.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Sub-tenon injection group (Experimental): In total twenty five subjects will be treated by injecting UMSCs in sub-tenon space of eye.
  Interventions: Biological: Injection of stem cells in sub-tenon space of eye for the management of retinitis pigmentosa
- Suprachoroidal injection group (Experimental): A total of twenty five subjects will be treated by suprachoroidal injection of UMSCs.
  Interventions: Biological: Injection of stem cells in suprachoroidal space of eye for the management of Retinitis Pigmentosa

INTERVENTIONS:
Biological: Injection of stem cells in sub-tenon space of eye for the management of retinitis pigmentosa — Cultured stem cells will be injected in the sub-tenon space of eye and patients will be monitored and evaluated for outer retinal thickness, early treatment of diabetic retinopathy study visual acuity, visual field sensitivity, fundus photography, amplitudes of multifocal electroretinogram and implicit times of multifocal electroretinogram at baseline (day 0) and days 30, 60, 90, 180, 270 and 360.
  Arms: Sub-tenon injection group
Biological: Injection of stem cells in suprachoroidal space of eye for the management of Retinitis Pigmentosa — Cultured stem cells will be injected in the suprachoroidal space of eye and patients will be monitored and evaluated for outer retinal thickness, early treatment of diabetic retinopathy study visual acuity, visual field sensitivity, fundus photography, amplitudes of multifocal electroretinogram and implicit times of multifocal electroretinogram at baseline (day 0) and days 30, 60, 90, 180, 270 and 360.
  Arms: Suprachoroidal injection group

SUMMARY:
Retinitis pigmentosa (RP) is the most common hereditary retinal disorder (accounts for 20% of children attending blind schools in Pakistan) which causes degeneration of rod and cone photoreceptors. Rods and cones largely depend on the retinal pigment epithelium for their proper functioning. Various growth factors and their receptors are present in retinal epithelium and a number of genes are responsible for the production of these growth factors. Genetic mutation in any of these genes causes retinal degeneration by progressive loss of retinal pigment epithelium and photoreceptors. The disease initially starts with night blindness and leads to the loss of central vision and eventually total blindness. To date, there is no definitive cure for patients suffering from RP. Recently, stem cell based therapies have shown great promise for the management of RP. It is well documented that umbilical cord derived mesenchymal stem cells (UMSCs) have the ability to release various paracrine and immunomodulatory factors that are similar to those synthesized by retinal pigment epithelium. Multiple routes including systemic (intravenous) and localized (subretinal, intravitreal, suprachoroidal and sub-tenon) have been employed to administer UMSCs for the management of RP. It is important to note that deep sub-tenon region (space between the sclera and the conjunctiva) acts as both natural culture medium for cells and as immune privileged site because of avascularity of the region. It has been reported that the injection of UMSCs in sub-tenon space of human subjects have improved the visual acuity even after 1 year post-injection. In addition, the injection of UMSCs in suprachoroidal space enhances the entry of growth factors released by the cells into choroidal flow and maintain the constant growth factors secretion to the choroidal and retinal tissues. Limoli and colleagues were the first to report the suprachoroidal administration of cells being the safe mode of cell delivery with no complications. The present study is aimed to investigate the safety and therapeutic efficacy of UMSC injection employing two different routes (sub-tenon injection versus suprachoroidal injection) for the treatment of RP in human subjects.

DETAILED DESCRIPTION:
Isolation and characterization of human umbilical cord derived mesenchymal stem cells (UMSCs): The culturing and characterization of UMSCs will be performed as documented by Ali and colleagues. Briefly, human umbilical cord tissues along with informed consent forms will be collected from COVID-19- and hepatitis B, C virus-negative women with healthy pregnancies during the Cesarean Section surgery after completion of gestation period. The umbilical cord tissue will be transported in sterile 1x phosphate-buffered saline (PBS) containing penicillin and streptomycin on ice. In the biosafety cabinet, the cord will be washed with 4-5 changes of sterile 1x PBS and placed in a Petri plate with 15ml PBS. The cord will then gently scrap with a surgical blade to remove any dead cells. A 9 cm umbilical cord will be cut into three equal pieces and wash thoroughly to remove blood clots, umbilical cord arteries, and veins. Segments will be washed three times with PBS and minced. The minced pieces will be incubated in 17.5ml of collagenase solution (201 U/ml collagenase type I in serum-free DMEM-HG) in a 50ml conical tube for ~3 hrs in an incubator at 5% CO2, 95% humidity at 37oC. After ~3 hrs, the digested lysate will be passed through strainer and will be diluted three times with 1x PBS. Following centrifugation, the cells will be seeded into two T-25cm2 flasks and will be placed in an incubator at 5% CO2, 95% humidity at 37o C. The flasks will be fed with fresh media (DMEM-HG supplemented with 20% FBS and 1% antibiotic solution) every third day. At around day 18, cells will reach up to 85% confluency and will be transferred in two T-75cm2 flasks with media replaced at alternate days. UMSCs at P3 will be characterized using different specific antibodies. Cells at P3 will be employed for injection in RP patients.

ELIGIBILITY:
Inclusion Criteria:

* Patients who will be voluntarily participated for UMSCs injection for the treatment of RP.
* Patients who will be able to adhere to the study follow-up and protocol requirements.
* Individuals with age ranges from 18 years to 70 years will be included.
* Patients with best corrected visual acuity (BCVA) from 50 letters to 110 letters or <20/50 in the ETDRS chart testing (Topcon CC-100 XP, Japan).
* Mean deviation values ranging between -33.0 and - 5.0 dB with compass visual field analysis (threshold 24-2, Sita Standard, Stimulus 3-white).
* Diagnosis of any phenotypic or genotypic variation of RP, confirmed by clinical history, fundus appearance, visual field, electroretinogram and genetic mutation analysis.

Exclusion Criteria:

* Presence of cataracts or other media opacity that might affect the visual field, mean deviation, or electroretinogram recordings.
* Presence of another ocular disease except RP (i.e., uveitis, strabismus, glaucoma) that causes visual field and optic disc changes.
* Presence of any systemic disorder that may affect visual functions. This includes diabetes, neurological disorders, and uncontrolled systemic hypertension.
* Smokers will be excluded from the study.
* Individuals who underwent ocular surgery except cataract extraction will be considered as excluded.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 50 (Estimated)
Dates: Start 2021-02 (Estimated); Primary Completion 2022-05 (Estimated); Study Completion 2022-06 (Estimated)

PRIMARY OUTCOMES:
Evaluation of safety related adverse ocular events including immune response | Baseline to day 360
  No significant side effects in stem cell treated subjects
Ophthalmic examination for best-corrected visual acuity (BCVA) using early treatment of diabetic retinopathy study (ETDRS) chart | Baseline to day 360
  Change in best corrected visual acuity (BCVA)

SECONDARY OUTCOMES:
Measurement of electrical activity/function of retina using Electroretinography (ERG) test | Baseline to day 360
  Change in electrical response/function of various cell types of retina
Evaluation of outer retinal thickness using Optical Coherence Tomography (OCT) imaging test | Baseline to day 360
  Alteration in retinal thickness
Examination of retinal damage by Fundus Photography | Baseline to day 360
  Change in retinal Fundus image
Evaluation of visual field sensitivity using perimeter | Baseline to day 360
  Change in visual field sensitivity

CONTACTS AND LOCATIONS:
Overall Officials: Sheikh Riazuddin, PhD, Principal Investigator — Jinnah Burn & Reconstructive Surgery Center, Lahore; Zaheer-ud-Din A Qazi, consultant, Principal Investigator — The Layton Rahmatullah Benevolent Trust (LRBT)
Locations (1):
- Stem Cell laboratory, Jinnah Burn & Reconstructive Surgery Centre, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kahraman NS, Oner A. Umbilical cord derived mesenchymal stem cell implantation in retinitis pigmentosa: a 6-month follow-up results of a phase 3 trial. Int J Ophthalmol. 2020 Sep 18;13(9):1423-1429. doi: 10.18240/ijo.2020.09.14. eCollection 2020. PMID 32953582
- [Background] Azam M, Collin RW, Malik A, Khan MI, Shah ST, Shah AA, Hussain A, Sadeque A, Arimadyo K, Ajmal M, Azam A, Qureshi N, Bokhari H, Strom TM, Cremers FP, Qamar R, den Hollander AI. Identification of novel mutations in Pakistani families with autosomal recessive retinitis pigmentosa. Arch Ophthalmol. 2011 Oct;129(10):1377-8. doi: 10.1001/archophthalmol.2011.290. No abstract available. PMID 21987686
- [Background] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly derived mesenchymal stem cells: preliminary clinical results. Stem Cell Res Ther. 2020 Jan 13;11(1):25. doi: 10.1186/s13287-020-1549-6. PMID 31931872
- [Background] Ozmert E, Arslan U. Management of retinitis pigmentosa by Wharton's jelly-derived mesenchymal stem cells: prospective analysis of 1-year results. Stem Cell Res Ther. 2020 Aug 12;11(1):353. doi: 10.1186/s13287-020-01870-w. PMID 32787913
- [Background] Limoli PG, Vingolo EM, Morales MU, Nebbioso M, Limoli C. Preliminary study on electrophysiological changes after cellular autograft in age-related macular degeneration. Medicine (Baltimore). 2014 Dec;93(29):e355. doi: 10.1097/MD.0000000000000355. PMID 25546695
- [Background] Ali M, Mehmood A, Tarar MN, Nawaz Z, Riazuddin SA, Khan A, Riazuddin S. Efficacy of intravenous infusions of UC-derived MSCs for the treatment of COVID-19: A structured summary of a phase II double blinded, randomized controlled clinical trial. Preprint from Research Square, 28 Oct 2020. DOI: 10.21203/rs.3.rs-92995/v2